CLINICAL TRIAL: NCT02384564
Title: A Randomized Comparison of the King Vision Video Laryngoscope aBlade vs. Direct Laryngoscopy in Children
Brief Title: King Vision Video Laryngoscope aBlade vs. Direct Laryngoscopy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator; M.D., Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB 2015-304
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Tracheal Intubation
Keywords: Laryngoscopy; Video Laryngoscopy; Tracheal intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambu King Vision Video Laryngoscope aBlade System (Experimental): The trachea will be intubated using the Ambu King Vision Video Laryngoscope with the appropriate sized blade (size 1 or 2) based on manufacturer guidelines and clinical judgement.
  Interventions: Device: Ambu King Vision Video Laryngoscope aBlade
- Direct Laryngoscope (Active Comparator): The trachea will be intubated via direct laryngoscopy using a traditional straight blade laryngoscope, with appropriately sized blade based on manufacturer guidelines and clinical judgement.
  Interventions: Device: Direct Laryngoscopy via Miller Straight Blade

INTERVENTIONS:
Device: Ambu King Vision Video Laryngoscope aBlade — At time of tracheal intubation, the subject will be intubated using the Ambu King Vision Video Laryngoscope with the appropriately sized Ambu aBlade System based on manufacturer guidelines and clinical judgement. The first attempt to successful intubation will be assessed. The Cormack Lehane and Percentage of Glottic Opening scores will be recorded via direct vision. Information on subsequent attempts, time to successful intubation, and ease of tracheal tube insertion will be assessed.
  Other Names: King Vision Video Laryngoscope
  Arms: Ambu King Vision Video Laryngoscope aBlade System
Device: Direct Laryngoscopy via Miller Straight Blade — At time of tracheal intubation, the subject will be intubated via direct laryngoscopy using a straight laryngoscope blade, based on manufacturer guidelines and clinical judgement. The first attempt to successful intubation will be assessed. The Cormack Lehane and Percentage of Glottic Opening scores will be recorded via direct vision. Information on subsequent attempts, time to successful intubation, and ease of tracheal tube insertion will be assessed.
  Other Names: Miller Blade, Wisconsin blade, Straight blade
  Arms: Direct Laryngoscope

SUMMARY:
The purpose of this study is to determine whether there is a clinically relevant difference in first attempt success rates between the Ambu King Vision Video Laryngoscope and Direct Laryngoscopy in Children.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to compare whether there is a clinically relevant difference in the rate of first attempt successful intubation between the Ambu King Vision Video Laryngoscope and direct laryngoscopy using the Miller Blade Laryngoscope. Other parameters of clinical relevance such as grade of laryngeal view, percentage of glottic opening, number of insertion attempts, time for successful tracheal intubation, and complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I-III classified patients
* Patients undergoing procedure where an endotracheal tube would be normally utilized

Exclusion Criteria:

* Children with expected difficult airways
* Coagulopathy

Ages: 1 Day to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
First Attempt Success Rate of Tracheal Intubation | Assessed intraoperatively at time of intubation
  An attempt at tracheal intubation will be defined as entry of the device into the patient's mouth without the need to remove the device once entered and securing the airway.

SECONDARY OUTCOMES:
Grades of Laryngeal View | Assessed intraoperatively at time of intubation
  Cormack Lehane (1-4) and percentage of glottic opening (POGO) (%) will be recorded after insertion of the laryngoscope.
Time to Successful Intubation | Assessed intraoperatively at time of intubation
  The time to intubation will be measured (seconds) to measure the time to intubation of the successful attempt.
Intraoperative Complications | Assessed intraoperatively for the duration of the surgery
  Airway/device related complications including, laryngospasm, bronchospasm, regurgitation/aspiration, oxygen desaturation, will be measured.
Postoperative Complications | Outcome measure will be assessed postoperatively in the immediate phase 1 recovery unit for an average of 1 hour.
  Airway/device related complications including sore throat, hoarseness, persistent coughing, stridor, and others will be measured during the post-operative period.
Ease of Endotracheal Tube Passage | Assessed intraoperatively at time of intubation
  The ease of tracheal tube passage will be measured following tracheal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: narasimhan jagannathan, MD, Principal Investigator — Ann & Robert Lurie Children's Hospital of Chicago

REFERENCES:
- [Background] Levitan RM, Heitz JW, Sweeney M, Cooper RM. The complexities of tracheal intubation with direct laryngoscopy and alternative intubation devices. Ann Emerg Med. 2011 Mar;57(3):240-7. doi: 10.1016/j.annemergmed.2010.05.035. Epub 2010 Jul 31. PMID 20674088
- [Background] Theiler L, Hermann K, Schoettker P, Savoldelli G, Urwyler N, Kleine-Brueggeney M, Arheart KL, Greif R. SWIVIT--Swiss video-intubation trial evaluating video-laryngoscopes in a simulated difficult airway scenario: study protocol for a multicenter prospective randomized controlled trial in Switzerland. Trials. 2013 Apr 4;14:94. doi: 10.1186/1745-6215-14-94. PMID 23556410
- [Background] Murphy LD, Kovacs GJ, Reardon PM, Law JA. Comparison of the king vision video laryngoscope with the macintosh laryngoscope. J Emerg Med. 2014 Aug;47(2):239-46. doi: 10.1016/j.jemermed.2014.02.008. Epub 2014 Apr 16. PMID 24742495
- [Background] Akihisa Y, Maruyama K, Koyama Y, Yamada R, Ogura A, Andoh T. Comparison of intubation performance between the King Vision and Macintosh laryngoscopes in novice personnel: a randomized, crossover manikin study. J Anesth. 2014 Feb;28(1):51-7. doi: 10.1007/s00540-013-1666-9. Epub 2013 Jun 30. PMID 23812581